CLINICAL TRIAL: NCT00249938
Title: Evaluation of Plant Sterol and Placebo on Low-density Lipoprotein Concentrations in Hyperlipidemic Patients Treated With Combination Statin and Colesevelam Therapy.
Brief Title: Evaluation of Combination Cholesterol Treatments in Patients With High Cholesterol.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-0823
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Hyperlipidemia; Dyslipidemia
Keywords: Antilipemic agents; hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias; Dyslipidemias | interventions — Colesevelam Hydrochloride

INTERVENTIONS:
Drug: Minute Maid Heart Wise orange juice
Drug: Welchol

SUMMARY:
The purpose of this study is to see if combination therapy with a "statin" medication and two additional agents that work differently than "statin" medications can further lower the so-called "bad cholesterol." One therapy is a prescription drug approved by the Food and Drug Administration to treat high cholesterol (Welchol). The other therapy is Minute Maid Heart Wise orange juice. This study juice is available in supermarkets and contains plant sterols that have been shown to lower cholesterol.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is the primary cause of morbidity and mortality in the United States. Lowering LDL cholesterol in both patients with and without CHD reduces coronary events and death. Statin medications are the primary mechanism of lowering LDL cholesterol, but some patients do not reach their goal LDL with maximum tolerated statin doses and must utilize combination therapy to further lower cholesterol. Additionally, some patients prefer to utilize "natural" mechanisms to lower cholesterol. This prospective, double-blinded, randomized study will compare plant sterol (natural cholesterol treatment) with placebo in patients treated with combination statin and colesevelam therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high cholesterol being treated with a statin
* LDL cholesterol greater than 100
* Ability to swallow large tablets

Exclusion Criteria:

* Diabetes
* Use of other medications to treat high cholesterol
* History of liver disease

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-03; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol

SECONDARY OUTCOMES:
Triglycerides, HDL cholesterol, total cholesterol, C-reactive protein, Apolipoprotein B

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Linnebur, Pharm.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver and Health Sciences Center, Denver, Colorado, United States